CLINICAL TRIAL: NCT05056207
Title: PREVENT: PeRomEter Visualization to ENd Treatment-related Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017-0639; NCI-2019-02478 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort I (patients receiving annual lymphedema screening) (Other): We will retrospectively retrieve information on patients who previously underwent preoperative perometer lymphedema screening during the past year who were treated definitively for their breast cancer with an ALND, and for whom no follow-up postoperative lymphedema screening was done.
  Interventions: Other: Cohort I (patients receiving annual lymphedema screening
- Cohort II (patients followed intensively for lymphedema) (Other): We will prospectively follow a cohort of 279 patients who have recently undergone ALND in this upcoming year with intensive lymphedema screening.
  Interventions: Other: Cohort II (patients followed intensively for lymphedema)

INTERVENTIONS:
Other: Cohort I (patients receiving annual lymphedema screening — patientns who previously underwent preoperative perometer lymphedema screening
  Arms: Cohort I (patients receiving annual lymphedema screening)
Other: Cohort II (patients followed intensively for lymphedema) — patients who have recently undergone ALND
  Arms: Cohort II (patients followed intensively for lymphedema)

SUMMARY:
This research study is to learn about breast cancer patients' opinions about screening for lymphedema (a side effect of breast cancer treatment in which the arm can become heavy, painful, and/or swollen) and their satisfaction with the lymphedema screening program.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the effectiveness of prospective, intensive lymphedema screening in the postoperative setting using a perometer for reducing the cumulative incidence of grade lymphedema among breast cancer patients after ALND compared to routine screening. Secondary Objectives:
* To estimate the direct costs associated with the Lymphedema Screening Initiative
* To determine the association of the Initiative on patient productivity
* To determine patient satisfaction with the Lymphedema Initiative in the context of their cancer care
* To determine patient understanding of lymphedema-associated symptoms
* To determine patient self-reported compliance with treatments and measures to prevent lymphedema
* To determine the incidence of breast cancer-related lymphedema among a cohort of breast cancer patients treated with ALND To analyze clinical and pathological features associated with the development of lymphedema

ELIGIBILITY:
Inclusion Criteria:

a Cohort A:

* Breast cancer patients with a baseline (preoperative perometer measurements) who have undergone axillary lymph node dissection
* English speaker
* Patients who participate in Cohort A will be eligible for enrollment in Cohort

b Cohort I:

* Breast cancer patients who have undergone axillary lymph node dissection who have a clinic visit in the Nellie B. Connally Breast Center approximately 12 months (+/- 4 months) following axillary lymph node dissection
* English speaker

c Cohort II:

* Breast cancer patients who have undergone axillary lymph node dissection who are having a follow-up visit in the Nellie B. Connally Breast Center within 0-6 months following surgery who intend to continue follow-up care at MD Anderson
* English speaker

Exclusion Criteria:

Inability to complete a self-administered questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
To establish the effectiveness of prospective, intensive lymphedema screening in the postoperative setting using a perometer. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simona Shaitelman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org